CLINICAL TRIAL: NCT04458961
Title: MIKROBE Management of Infected Knee Replacements-Obtaining Best Evidence A Feasibility Study for a Randomised Controlled Trial of One-stage or Two-stage Surgery for Prosthetic Knee Infection
Brief Title: MIKROBE Management of Infected Knee Replacements-Obtaining Best Evidence
Acronym: MIKROBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); Nuffield Orthopaedic Centre NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 272334
Record Dates: First submitted 2020-06-05; First posted 2020-07-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Arthropathy; Arthropathy Related to Infection; Arthropathy of Knee Joint; One-stage; Two-stage; Infection; Prosthetic joint infection
MeSH Terms: conditions — Joint Diseases; Infections

STUDY DESIGN:
Masking Description: Blinding of participants and trial personnel will not be possible due to the nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-stage (Active Comparator)
  Interventions: Procedure: One-stage
- Two-stage (Active Comparator)
  Interventions: Procedure: Two-stage

INTERVENTIONS:
Procedure: One-stage — A one-stage revision operation involves one operation to remove the joint, thoroughly cleaning the infected area and then implanting a new joint immediately.
  Arms: One-stage
Procedure: Two-stage — A two-stage revision operation involves two operations: the joint is removed in one operation, a temporary spacer device is inserted, then the infection is treated with antibiotics, and then a new joint is implanted in a second operation.
  Arms: Two-stage

SUMMARY:
Following a prosthetic knee joint infection, two types of operative approach can be undertaken to treat the infection: a one-stage or two-stage revision operation. Both approaches are widely used and are good at treating infection but we don't know which has the best long-term outcomes for patients. This trial aims to assess the feasibility of conducting a randomised controlled trial to evaluate whether treating a prosthetic knee infection with one-stage revision surgery gives a better outcome than two-stage revision surgery in terms of patient function and pain, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adults with prosthetic knee infection suitable for either one-stage or two-stage revision surgery
* Intra-operatively, all cases must have adequate soft-tissue coverage post debridement to allow single or two stage revision surgery.
* Case meets the International Consensus Meeting criteria for infection
* Patients having had a Debridement, Anti-biotic and Implant Retained procedure previously or washout/biopsy only of an infected TKR are suitable

Exclusion Criteria:

* Unable or unwilling to undergo either treatment
* Lacking capacity to consent to research
* Refusal to consent to study for any reason
* Re-revision of prosthetic knee infection if first revision was for infection
* Presence of tuberculosis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Ease of recruitment of participants | 20 months
  Number of recruits compared to the number of potential participants.

SECONDARY OUTCOMES:
Explaining the study | 20 months
  Assessment of the process of explaining the study (explanation/recruitment/randomisation) between patients and surgeons via qualitative analysis of audio recording of pre-operative discussions about entering the study.
Reasons for non-participation | 20 months
  Qualitative analysis of semi-structured interviews with those patients who declined to participate in the trial.
Patient experience | 2 weeks after surgery
  Experience and acceptability of the process of recruitment, randomisation and study participation via qualitative analysis of semi-structured interview.
Surgeon experience | 20 months
  Experience of the process of recruitment, randomisation and study participation including thoughts about trial design via qualitative analysis of semi-structured interview after each patient surgery and at the end of the trial.
Protocol adherence | 20 months
  Assessment of any deviations or violations to protocol that occur during the trial.
Healthcare resource utilisation | 20 months
  Patient-reported questionnaire assessing heath and social resource use through an adapted questionnaire of the Client Service Receipt Inventory (CSRI) at 3 and 6 months post-operatively
Comparison of two sites | 20 months
  Recruitment and attrition rates at the two sites
Knee injury and Osteoarthritis Outcome Score (KOOS) outcome and completion rates | 20 months
  Patient-reported questionnaire assessing short-term and long-term symptoms and function in patients with knee injury to be administered pre-, 3 months and 6 months post-operatively
Oxford Knee Score (OKS) outcome and completion rates | 20 months
  Patient-reported questionnaire assessing function and pain after total knee replacement surgery to be administered pre-, 3 months and 6 months post-operatively
EQ-5D-5L outcome and completion rates | 20 months
  Patient-reported questionnaire assessing health-related quality of life to be administered pre-, 3 months and 6 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Toms, FRCS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Princess Elizabeth Orthopaedic Centre, Royal Devon and Exeter NHS Trust (RD&E NHSFT), Exeter, Devon
  - Nuffiels Orthopaedic Centre (NOC), Oxford

REFERENCES:
- [Derived] Terry R, Dean S, Hourigan P, Waterson HB, Wylde V, Carpenter N, Whale B, Powell RJ, Tarrant P, Medina-Lara A, Alvand A, Toms AD. MIKROBE: a feasibility study for a randomised controlled trial of one-stage or two-stage surgery for prosthetic knee infection. Pilot Feasibility Stud. 2025 Apr 16;11(1):49. doi: 10.1186/s40814-025-01634-4. PMID 40241215